CLINICAL TRIAL: NCT06655051
Title: Efficacy and Safety of Single Plastic Stent Compared With Fully Covered Self-Expanding Metal Stent on Benign Biliary Stricture Secondary to Chronic Pancreatitis: A Single Center，Prospective，Non-inferiority, Open Label, Randomized, Controlled Trial
Brief Title: Single Plastic Stent Vs. Fully Covered Self-Expanding Metal Stent on Benign Biliary Stricture Secondary to Chronic Pancreatitis
Acronym: ESSENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESSENCE202405
Record Dates: First submitted 2024-10-19; First posted 2024-10-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pancreatitis; Benign Biliary Stricture
Keywords: chronic pancreatitis; benign biliary stricture; ERCP; ERBD; stent
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fully covered self-expanding metal stent (Active Comparator): A single biliary fcSEMS will be placed under ERCP. During stenting period , if symptoms of biliary obstruction occur due to stent occlusion or migration, ERCP replacement or implantation of a new stent should be performed according to the condition. After 6 months of stenting, imaging evaluation will be performed. ERCP is not needed if the stent undergoes spontaneous complete distal migration and the patient is asymptomatic and has normal liver function. If the stent is visible, ERCP will be performed to remove the stent and the stricture will be evaluated. If stricture persists after 6 months of stenting, a follow-up treatment plan should be developed through multidisciplinary discussion. One month after ERCP, complications will be followed up by telephone. Follow-up after biliary stent removal will be conducted to inquire about symptoms, signs and liver function test results, and to evaluate the recurrence of biliary stricture.
  Interventions: Device: endoscopic retrograde biliary drainage ( fully covered self-expanding metal stent)
- single plastic stent (Experimental): A single biliary plastic stent will be placed under ERCP. During stenting period , if symptoms of biliary obstruction occur due to stent occlusion or migration, ERCP replacement or implantation of a new stent should be performed according to the condition. After 6 months of stenting, imaging evaluation will be performed. ERCP is not needed if the stent undergoes spontaneous complete distal migration and the patient is asymptomatic and has normal liver function. If the stent is visible, ERCP will be performed to remove the stent and the stricture will be evaluated. If stricture persists after 6 months of stenting, a follow-up treatment plan should be developed through multidisciplinary discussion. One month after ERCP, complications will be followed up by telephone. Follow-up after biliary stent removal will be conducted to inquire about symptoms, signs and liver function test results, and to evaluate the recurrence of biliary stricture.
  Interventions: Device: endoscopic retrograde biliary drainage (single plastic stent)

INTERVENTIONS:
Device: endoscopic retrograde biliary drainage (single plastic stent) — Participants will undergo ERCP. A flexible tube is inserted into the duodenum, crossing the sphincter of Oddi to access the biliary system. And the location, diameter, and length of biliary stricture will be evaluated by injection of contrast media. A single plastic stent is then placed across the biliary stricture, allowing the bile duct to resume drainage. The participants will be observed closely after ERCP and record complications. Imaging evaluation will be conducted 6 months after stenting to confirm spontaneous passage of the biliary duct stent, and the stent will be removed via ERCP if it is still in place.
  Arms: single plastic stent
Device: endoscopic retrograde biliary drainage ( fully covered self-expanding metal stent) — Participants will undergo ERCP. A flexible tube is inserted into the duodenum, crossing the sphincter of Oddi to access the biliary system. And the location, diameter, and length of biliary stricture will be evaluated by injection of contrast media. A fully covered self-expanding metal stent is then placed across the biliary stricture, allowing the bile duct to resume drainage. The participants will be observed closely after ERCP and record complications. Imaging evaluation will be conducted 6 months after stenting to confirm spontaneous passage of the biliary duct stent, and the stent will be removed via ERCP if it is still in place.
  Arms: Fully covered self-expanding metal stent

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of a single plastic stent versus a fully covered self-expanded metal stent in relieving benign biliary stricture secondary to chronic pancreatitis. The main questions it aims to answer is:

Whether the efficacy of a single plastic stent is non-inferior to that of a fully covered metal stent in patients with benign biliary stricture secondary to chronic pancreatitis？

Participants will be randomly assigned to receive either a single plastic stent (SPS) placement or fully covered self-expanded metal stent placement treatment for 6 months, and they will be followed up for 18 months.

DETAILED DESCRIPTION:
Although a number of previous studies have shown that the drainage and dilation effect of a single plastic stent is limited for benign biliary stricture (BBS) secondary to chronic pancreatitis (CP), the poor management of CP itself in most studies may explain the unsatisfactory efficacy of a single biliary plastic stent in relieving CP secondary BBS. Investigators believe that the effective management of CP is an important step to solve the BBS secondary to CP, especially the effective removal of pancreatic duct stones, the relief of pancreatic duct obstruction and the maintenance of pancreatic duct patency. Previous data showed that in CP patients treated with ESWL combined with ERCP, 72.4% could achieve complete removal of main pancreatic duct stones and 90.8% could achieve successful endoscopic decompression. Under the premise of effectively removing the stones of the main pancreatic duct at the head of the pancreas and maintaining the patency of the pancreatic duct, using a single plastic stent for stent drainage of BBS is effective, and a single plastic stent has potential advantages such as lower stent displacement rate and cheaper. Therefore, investigators design a single-center, prospective, open-label, randomized controlled, non-inferiority trial to compare the effectiveness, safety, and cost-effectiveness of a single plastic stent and fcSEMS for the removal of CP secondary BBS under the premise that the primary disease, i.e. CP itself, was effectively managed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. Patients diagnosed with CP;
3. Symptomatic biliary stricture documented at time of enrollment for naïve stricture or at the time of prior plastic stent placement in strictures that had 1 prior plastic stent inserted: cholangitis, and/or an increase in total bilirubin or alkaline phosphatase levels(> 2 times the upper limit of normal) for more than 4 weeks;
4. Confirmation of bile duct stricture by imaging assessment.

Exclusion Criteria:

1. Prior plastic stenting exceeding six months or any metal stenting;
2. Incomplete removal of stones from the main pancreatic duct located in the head of the pancreas during ERCP procedures;
3. Biliary stricture of benign etiology other than chronic pancreatitis;
4. Developing obstructive biliary symptoms associated with an attack of acute pancreatitis;
5. Stricture within 2 cm of common bile duct bifurcation;
6. Biliary stricture of malignant etiology;
7. Patients with acute or chronic hepatitis, cirrhosis, primary sclerosing cholangitis, congenital biliary malformations or biliary fistula;
8. Symptomatic duodenal stenosis (with gastric stasis);
9. Subjects for whom endoscopic techniques are contraindicated;
10. Pregnancy, incarceration;
11. Life expectancy < 1 year;
12. Other conditions that inappropriate to participant in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term stricture resolution | 2 years after enrollment
  Stricture resolution assessed at the time of final stent removal as well as the absence of objective findings of stricture recurrence during the 18 months, post-stenting follow-up period.

SECONDARY OUTCOMES:
Early clinical success | 6 months after enrollment
  Stricture resolution at the time all stent is removed. If there is a persistent stricture after 6 months of stent therapy in either group, the patient will be classified as a clinical failure.
Technical success | 6 months after enrollment
  The completion of the initial and each follow-up ERCP, including stent deployment and removal.
Adverse events related to the device or procedure | 2 years after enrollment
  Device or procedure related adverse events from the initial stent placement procedure to the 2 year follow-up.
Length of stent placement and removal procedures | 6 months after enrollment
  Length of stent placement procedures and stent removal procedures.
Number of ERCP procedures after Initial stent placement. | 6 months after enrollment
  The number of endoscopic retrograde cholangiopancreatography (ERCP) procedures after initial stent placement.
Number of stents placed | 6 months after enrollment
  The total number of stents placed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Study Chair — Changhai Hospital; Liang-Hao Hu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital Clinical Research Ward, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramchandani M, Pal P, Costamagna G. Management of Benign Biliary Stricture in Chronic Pancreatitis. Gastrointest Endosc Clin N Am. 2023 Oct;33(4):831-844. doi: 10.1016/j.giec.2023.04.002. Epub 2023 May 11. PMID 37709414
- [Background] Dumonceau JM, Delhaye M, Tringali A, Arvanitakis M, Sanchez-Yague A, Vaysse T, Aithal GP, Anderloni A, Bruno M, Cantu P, Deviere J, Dominguez-Munoz JE, Lekkerkerker S, Poley JW, Ramchandani M, Reddy N, van Hooft JE. Endoscopic treatment of chronic pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Updated August 2018. Endoscopy. 2019 Feb;51(2):179-193. doi: 10.1055/a-0822-0832. Epub 2019 Jan 17. PMID 30654394
- [Background] Deviere J, Nageshwar Reddy D, Puspok A, Ponchon T, Bruno MJ, Bourke MJ, Neuhaus H, Roy A, Gonzalez-Huix Llado F, Barkun AN, Kortan PP, Navarrete C, Peetermans J, Blero D, Lakhtakia S, Dolak W, Lepilliez V, Poley JW, Tringali A, Costamagna G; Benign Biliary Stenoses Working Group. Successful management of benign biliary strictures with fully covered self-expanding metal stents. Gastroenterology. 2014 Aug;147(2):385-95; quiz e15. doi: 10.1053/j.gastro.2014.04.043. Epub 2014 May 4. PMID 24801350
- [Background] Haapamaki C, Kylanpaa L, Udd M, Lindstrom O, Gronroos J, Saarela A, Mustonen H, Halttunen J. Randomized multicenter study of multiple plastic stents vs. covered self-expandable metallic stent in the treatment of biliary stricture in chronic pancreatitis. Endoscopy. 2015 Jul;47(7):605-10. doi: 10.1055/s-0034-1391331. Epub 2015 Jan 15. PMID 25590182
- [Background] Cote GA, Slivka A, Tarnasky P, Mullady DK, Elmunzer BJ, Elta G, Fogel E, Lehman G, McHenry L, Romagnuolo J, Menon S, Siddiqui UD, Watkins J, Lynch S, Denski C, Xu H, Sherman S. Effect of Covered Metallic Stents Compared With Plastic Stents on Benign Biliary Stricture Resolution: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1250-7. doi: 10.1001/jama.2016.2619. PMID 27002446
- [Background] Ramchandani M, Lakhtakia S, Costamagna G, Tringali A, Puspoek A, Tribl B, Dolak W, Deviere J, Arvanitakis M, van der Merwe S, Laleman W, Ponchon T, Lepilliez V, Gabbrielli A, Bernardoni L, Bruno MJ, Poley JW, Arnelo U, Lau J, Roy A, Bourke M, Kaffes A, Neuhaus H, Peetermans J, Rousseau M, Reddy DN. Fully Covered Self-Expanding Metal Stent vs Multiple Plastic Stents to Treat Benign Biliary Strictures Secondary to Chronic Pancreatitis: A Multicenter Randomized Trial. Gastroenterology. 2021 Jul;161(1):185-195. doi: 10.1053/j.gastro.2021.03.015. Epub 2021 Mar 17. PMID 33741314